CLINICAL TRIAL: NCT04206072
Title: A Phase II/III, Open-Label, Randomised Study to Assess the Safety and Efficacy of D-0316 Versus Icotinib as First Line Treatment in Patients With EGFR Sensitising Mutation, Locally Advanced or Metastatic NSCLC
Brief Title: D-0316 Versus Icotinib in Patients With Locally Advanced or Metastatic EGFR Sensitising Mutation Positive NSCLC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBIO-103
Record Dates: First submitted 2019-12-10; First posted 2019-12-20 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Non-Small Cell Lung Cancer; EGFR Gene Mutation
Keywords: D-0316; EGFR mutated NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- D-0316 (Experimental): D-0316 (75 mg or 100 mg orally, once daily), in accordance with the randomization schedule.
  Interventions: Drug: D-0316 Capsule
- Icotinib (Active Comparator): Icotinib (125 mg orally, three times daily), in accordance with the randomization schedule.
  Interventions: Drug: Icotinib Hydrochloride Tablets

INTERVENTIONS:
Drug: D-0316 Capsule — The initial dose of D-0316 is 75 mg orally once daily (QD) for one cycle, and then increased to 100 mg orally QD in the absence of CTCAE grade ≥ 2 headache or thrombocytopenia during the first cycle, otherwise maintained to 75 mg orally QD until disease progression or meet the discontinuation criteria. A cycle of treatment is defined as 21 days of once daily treatment.
  Following objective disease progression according to RECIST 1.1, as per investigator assessment, patients who were confirmed T790M mutation positive may have the option to continuously receive D-0316.
  Arms: D-0316
Drug: Icotinib Hydrochloride Tablets — Icotinib (125 mg three times daily, orally), treatment should continue until disease progression or meet the withdrawal criteria. A cycle of treatment is defined as 21 days of three times daily treatment.
  Following objective disease progression according to RECIST 1.1, as per investigator assessment, patients who were randomized to Icotinib arm and confirmed T790M mutation positive have the option to receive D-0316 (crossover to active D-0316).
  Other Names: Conmana
  Arms: Icotinib

SUMMARY:
To assess the efficacy and safety of D-0316 versus Icotinib, a standard of care epidermal growth factor receptor tyrosine kinase inhibitor (EGFR-TKI), in patients with locally advanced or Metastatic Non Small Cell Lung Cancer (NSCLC).

DETAILED DESCRIPTION:
This is a Phase II/III, open-label, randomised study assessing the efficacy and safety of D-0316 (70 mg once daily for 21 days, then increased to 100 mg once daily, orally) versus Icotinib (125 mg three times daily, orally) in patients with locally advanced or metastatic NSCLC that is known to be EGFR sensitising mutation (EGFRm) positive, treatment-naive and eligible for first-line treatment with an EGFR-TKI.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older.
* Pathologically confirmed adenocarcinoma of the lung, with locally advanced or metastatic disease and not amenable to curative surgery or radiotherapy (stage IIIB, IIIC or IV disease based on the eighth edition of the American Joint Committee on Cancer (AJCC) TNM classification). Patients with mixed histology are eligible if adenocarcinoma is the predominant histology.
* Patients must be treatment-naive for locally advanced or metastatic NSCLC and eligible to receive first-line treatment with icotinib. Prior adjuvant and neo-adjuvant therapy (except for EGFR-TKI) is permitted if have been completed at least 6 months prior to initiation of study drug.
* The tumour tissues harbour one of the two common EGFR mutations known to be associated with EGFR-TKI sensitivity (Ex19del, L858R), either alone or in combination with other EGFR mutations, assessed by central laboratory.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1
* Predicted survival ≥ 3 months
* At least 1 measurable tumor lesion as per RECIST v1.1
* Agree to use effective contraception during the study period and for at least 3 months after completion of the study treatment
* Provision of informed consent prior to any study procedure.

Exclusion Criteria:

* Evidence of any concurrent or history of malignancy (except for clinically cured in situ cervix carcinoma, basal cell or squamous epithelial skin cancer, thyroid papillary carcinoma).
* Prior treatment with EGFR-TKI.
* Prior treatment with any systemic anti-cancer therapy for locally advanced or metastatic NSCLC including chemotherapy, biological therapy, immunotherapy, and etc.
* Previous therapeutic clinical trial with 4 week of the first dose of study drug.
* Previous traditional chinese medicine with an anti-cancer indication within 2 weeks of the first dose of study drug.
* Previous major surgery (except for tooth extraction) within 4 weeks of the first dose of study drug, planing to have major surgery during study.
* Symptoms or signs worsened within 2 weeks before screening.
* Any unresolved toxicities from prior treatment greater than NCI CTCAE v4.03 grade 2 or higher, with the exception of hair loss.
* Spinal cord compression, symptomatic or unstable central nervous system (CNS) metastases that require the use of steroids. Patients who have a stable CNS status for at least 4 weeks before treatment will be allowed to join the study.
* Any evidence of serious or uncontrolled systemic disease, including uncontrolled hypertension and active bleeding diatheses, or active infection including hepatitis B, hepatitis C, syphilis and human immunodeficiency virus (HIV).
* Clinically significant cardiovascular disease, such as mean resting corrected QT interval (QTcF) ≥470 msec (female) or ≥450 msec (male), obtained from 3 ECGs, or any clinically important abnormalities in rhythm, conduction, or morphology of resting ECG or left ventricular ejection fraction (LVEF) ≤ 50%, etc.
* Previous history of interstitial lung disease, drug-induced interstitial lung disease, history of radiation-induced pneumonia requiring hormone therapy, or clinical evidence of active interstitial lung disease.
* Presence of active gastrointestinal disease or other condition that would preclude the absorption, distribution, metabolism, or excretion of study drug.
* Patients currently receiving medications known to be potent inducers, sensitive substrate or potent inhibitor of cytochrome P450 (CYP) 3A4 (e.g. CYP3A4), CYP3A5, CYP2D6 and CYP2C8.
* Patients with a known allergy or delayed hypersensitivity reaction to study drug or its excipient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2019-12-24 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Median Progression Free Survival (PFS) assessed by IRC | From randomization to objective disease progression or death, whichever came first, assessed up to 20 months
  PFS is defined as the time from randomization until the date of objective disease progression or death by any cause, whichever occurs first. The primary endpoint of PFS was based on independent review committee (IRC) assessment.

SECONDARY OUTCOMES:
Median Progression Free Survival (PFS) assessed by Investigator | From randomization to objective disease progression or death, whichever came first, assessed up to 20 months
  PFS is defined as the time from randomization until the date of objective disease progression or death by any cause, whichever occurs first.
Objective Response Rate (ORR) | At baseline and every 6 weeks (±4 days) until disease progression, up to 20 months
  ORR is defined as the percentage (%) of participants with measurable disease with a best overall response of complete response (CR) or partial response (PR). ORR was based on investigator and IRC assessment.
Duration of Response (DoR) | At baseline and every 6 weeks (±4 days) until disease progression, up to 20 months
  DoR is defined as the time from the date of first documented response (CR or PR) until the date of documented progression or death in the absence of disease progression. DoR was based on both Investigator and IRC assessment.
Disease Control Rate (DCR) | At baseline and every 6 weeks (±4 days) until disease progression, up to 20 months
  DCR is defined as the percentage (%) of participants who had a best overall response (BOR) of CR, PR or Stable disease (SD) ≥6 weeks prior to any progressive disease (PD) event, assessed by investigator and IRC.
Overall Survival (OS) | From randomization to date of death from any cause, whichever came first, up to 36 months
  OS is defined as the time from randomization until the date of death due to any cause.
Intracranial ORR (iORR) | At baseline and every 6 weeks (±4 days) until disease progression, up to 20 months
  iORR is calculated as the ORR (CR+PR) of lesions in the brain for patients who have measurable disease in the brain at baseline. iORR was based on both Investigator and IRC assessment.
Intracranial PFS (iPFS) | From randomization to objective intracranial disease progression or death, whichever came first, up to 20 months
  iPFS is defined as time from randomization to intracranial disease progression or death due to any causes, assessed by investigator and IRC.
Adverse event (AE) | At baseline and every 3 weeks (±4 days) for the first 6 weeks, and then every 6 weeks (±4 days) until objective disease progression or meet other withdrawal criteria, up to 36 months
  AE is defined as any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study medication, whether or not considered related to the study medication. AEs are summarized by type, incidence, severity and relationship to study medication.

OTHER OUTCOMES:
Change From Baseline Scores on the functional assessment of cancer therapy - Lung (FACT-L) quality of life questionnaire | At baseline and every 6 weeks (±4 days) until disease progression, up to 20 months
  The FACT-L questionnaire consists of several major aspects of life (Physical, social/family, emotional, and functional well-being) as well as lung cancer subscale (symptoms, cognitive function, regret of smoking). Scores for item ranging from 0 (not at all) to 4 (very much).

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu, PHD, Principal Investigator — Shanghai Chest Hospital
Locations (2):
- China (2):
  - The First Affiliated Hospital of Medical School of Zhejiang University, Hangzhou, Zhejiang
  - Liuzhou Workers Hospital, Liuchow

REFERENCES:
- [Derived] Lu S, Zhou J, Jian H, Wu L, Cheng Y, Fan Y, Fang J, Chen G, Zhang Z, Lv D, Jiang L, Wu R, Jin X, Zhang X, Zhang J, Xie C, Sun G, Huang D, Cui J, Guo R, Han Z, Chen Z, Liang J, Zhuang W, Hu X, Zang A, Zhang Y, Cang S, Lan Y, Chen X, Liu L, Li X, Chen J, Ma R, Guo Y, Sun P, Tian P, Pan Y, Liu Z, Cao P, Ding L, Wang Y, Yuan X, Wu P. Befotertinib (D-0316) versus icotinib as first-line therapy for patients with EGFR-mutated locally advanced or metastatic non-small-cell lung cancer: a multicentre, open-label, randomised phase 3 study. Lancet Respir Med. 2023 Oct;11(10):905-915. doi: 10.1016/S2213-2600(23)00183-2. Epub 2023 May 24. PMID 37244266
- [Derived] Lu S, Zhang Y, Zhang G, Zhou J, Cang S, Cheng Y, Wu G, Cao P, Lv D, Jian H, Chen C, Jin X, Tian P, Wang K, Jiang G, Chen G, Chen Q, Zhao H, Ding C, Guo R, Sun G, Wang B, Jiang L, Liu Z, Fang J, Yang J, Zhuang W, Liu Y, Zhang J, Pan Y, Chen J, Yu Q, Zhao M, Cui J, Li D, Yi T, Yu Z, Yang Y, Zhang Y, Zhi X, Huang Y, Wu R, Chen L, Zang A, Cao L, Li Q, Li X, Song Y, Wang D, Zhang S, Ding L, Zhang L, Yuan X, Yao L, Shen Z. Efficacy and Safety of Befotertinib (D-0316) in Patients With EGFR T790M-Mutated NSCLC That Had Progressed After Prior EGFR Tyrosine Kinase Inhibitor Therapy: A Phase 2, Multicenter, Single-Arm, Open-Label Study. J Thorac Oncol. 2022 Oct;17(10):1192-1204. doi: 10.1016/j.jtho.2022.06.002. Epub 2022 Jun 18. PMID 35724798